CLINICAL TRIAL: NCT02577874
Title: A Comparison of European and Chinese Blood Sugar Responses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Small Changes (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: Chinese European study 2015
Record Dates: First submitted 2015-06-15; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chinese Subjects: 7 blood glucose tests taken over a two hour period
- European Subjects: 7 blood glucose tests taken over a two hour period

SUMMARY:
This study is designed to compare the responses to an oral glucose challenge between people of European and Chinese heritage (essential participants in the European arm must have tow European parents and likewise for the Chinese participants).

DETAILED DESCRIPTION:
100 participants (50 European and 50 Chinese) will attend a lab after an overnight fast and have a capillary finger-prick blood test to assess fasted blood glucose levels and then consume a 50 gram glucose solution. Blood test will be repeated at 15, 30, 45, 60, 90 and 120 minutes post consumption of the glucose solution. This test will be repeated on a spate occasion at least a week later than the first test. Participants will only take part in the experiment after singing informed consent and agreeing to take part in the study and after a medical screening questionnaire assessing that they are non-diabetic or haemophiliac or have blood born infections.

ELIGIBILITY:
Inclusion Criteria:

* European ethnicity
* Chinese ethnicity
* age 19-59 years

Exclusion Criteria:

* diabetics
* serious blood born infection
* haemophilia

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health adults, male and female between the ages of 19 and 59
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Blood sugar response measured by 7 finger prick blood samples | 2 hours
  7 finger prick blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam Univeristy Food and Nutrition laboratory, Sheffield, South Yorkshire, United Kingdom